CLINICAL TRIAL: NCT05308758
Title: Effect of Game-based High-Intensity Interval Training Program on the Executive Function of Children With ADHD: Protocol of A Randomized Controlled Trial
Brief Title: Effect of Game-based HIIT Program on the Executive Function of Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EdUHK 18603120
Record Dates: First submitted 2022-02-17; First posted 2022-04-04 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-05

CONDITIONS: Adhd Deficits in Attention Motor Control and Perception
Keywords: Special education need; Physical activity; fNIRS
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to treatment allocation because of the intervention nature. To avoid contamination between treatment groups, intervention deliverers will be provided with a list of students in the intervention program. Only those on the list can participate in the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GameHIIT intervention group (Experimental): In the GameHIIT group, a specially designed game-based training program with HIIT in nature will be delivered to the participants for 8 weeks.
  Interventions: Other: Game-based High-Intensity Interval Training
- GameSE intervention group (Active Comparator): In the GameSAE group, participants will attend a tailor-made game-based exercise training program. Similar to GameHIIT, the intervention will comprise 8 weeks of structured aerobic exercise sessions, lasting one hour on average in each session and up to twice per week.
  Interventions: Other: GameSAE
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Other: Game-based High-Intensity Interval Training — There will be two training sessions each week. In each training session, there will be four sets of training programs separated by 3 minutes of passive recovery in accordance with a previous study.Each set of activities will last for around 5 minutes; therefore, the total duration of each training session will be approximately 30 minutes. A small group size (4-6 children per group) will be adopted to facilitate individual supervision and adaption of the exercise program.
  Arms: GameHIIT intervention group
Other: GameSAE — Similar to GameHIIT, the intervention will comprise 8 weeks of structured aerobic exercise sessions, lasting one hour on average in each session and up to twice per week. Six to eight stations of multidimensional exercises will be set up for each session. Adopting the train-the-trainer (TTT) model, training will be provided by front-line healthcare providers or trained helpers. Children will be instructed to finish the exercises in all stations one after another in a predetermined order.
  Arms: GameSE intervention group

SUMMARY:
Background: Attention-deficit/hyperactivity disorder (ADHD) is a common developmental disorder in childhood, with a 5%-6% worldwide prevalence. Children with ADHD often demonstrate impaired executive function, which is closely related to the development of the commonly observed behavioral problems such as inattention, impaired inhibition, and hyperactivity. The purpose of this study is to examine whether a game-based high-intensity interval training (HIIT) program can improve the executive function of children with ADHD, compared with a traditional structured aerobic exercise program and a non-treatment control group.

Methods/design: A total of 42 children with ADHD will be recruited to participate in this three-arm school-based randomized controlled trial. An 8-week specially designed game-based HIIT (GameHIIT) program and a traditional game-based structured aerobic exercise (GameSAE) program will be delivered to those children randomly assigned to these two intervention groups, while the children in the control group will maintain their regular physical activity over the same period. A number of outcome measures including executive function, cerebral hemodynamic response, physical activity, physical fitness, and enjoyment and adherence to the intervention will be assessed for both groups at baseline (T0), immediately after the intervention period (T1), and after the follow-up period (T2).

Discussion: HIIT has recently emerged as a feasible and efficacious strategy for increasing physical health outcomes and cognitive function, including executive function, in healthy young people. However, research has yet to investigate whether the executive function of children with ADHD can be effectively enhanced through HIIT. If, as hypothesized, GameHIIT program improves outcomes for children with ADHD, the present research will inform the development of targeted exercise programs that can be more broadly used with this particular population.

Keywords: Special education need, Physical activity, fNIRS,

DETAILED DESCRIPTION:
There is strong evidence that regular physical activity (PA) is associated with a range of physical health benefits for school-age youth, including improvements in body composition, physical capacity, and overall health-related indicators (e.g., blood pressure, insulin resistance, lipid profile). Emerging evidence also suggests that PA and physical fitness have a positive effect on mental health, cognitive function, and academic performance. Executive functions are generally defined as "high-level cognitive processes" that manage other basic cognitive functions. They consist of functions such as planning, self-regulation, initiation and inhibition, and cognitive flexibility. These functions are believed to be important prerequisites for successful learning in preadolescent children, predict better health and wealth, and have been associated with a reduced likelihood of being convicted of a criminal offense. Several recent meta-analyses have suggested that PA may positively affect cognition and executive function in children. Despite the known benefits of an active lifestyle, more than half of Hong Kong's children and young people fail to follow the current physical activity recommendations, and trends show a decline in health-related physical fitness. Executive functions develop from early childhood and through adolescence into adulthood, with large developmental changes occurring during the elementary school years. Accordingly, effective interventions implemented early in life when the higher cortex is still developing, have the potential to elicit significant long-term improvements. Therefore, it is important to find effective strategies to promote the PA of children, so as to improve their executive function during their childhood.

Attention-deficit/hyperactivity disorder (ADHD) is a commonly diagnosed developmental disorder, with a 5.3% worldwide prevalence in children and adolescents. The most common symptoms include inattention, impulsivity, impaired inhibition, and hyperactivity. Also, young people with ADHD are often characterized by dysfunction in high-level cognitive functions such as executive function. This executive dysfunction may play an important role in the commonly observed behavioral problems in children with ADHD. There are a number of ways to treat ADHD, e.g., medication, psychotherapy, psychoeducation, neuro-feedback, behavior management, etc. Of these treatments, PA and exercise have emerged as effective strategies to manage ADHD given that neither are associated with negative side effects (see recent reviews. To summarize, although not always consistently, PA, especially moderate- to high-intensity aerobic exercise, may improve the emotion/mood, behavior, executive function, and some physical measures of children with ADHD. Acute aerobic exercise may have a positive effect on a variety of measures with a large effect size up to 1.26 in children with ADHD. Two studies have reported medium-to-large effects of acute exercise on executive function. Long-term exercise interventions have also been shown to benefit children with ADHD, with improvements in some measures showing a large effect size up to 0.96. However, these benefits have been mainly described as an improvement of behavioral and emotional problems. Several studies have reported that long-term 'mixed exercise programs' may have moderate to significant effects on several aspects of executive function (e.g., inhibition) and attention in children and adolescents with ADHD, but other studies did not report the same findings. Therefore, so far evidence-based suggestions regarding the optimal exercise for children with ADHD remain somewhat inconsistent.

Research into the relationship between PA and ADHD has generally involved mixed exercise programs at a low- to moderate-intensity; running and stationary cycling have been the most common exercise modes. Whether structured PA is effective for young people is yet to be examined. Children's habitual PA patterns are characterized by participation in games or "unpredictable" sports activities (e.g., football, basketball). Given that children's intrinsic motivation, or level of enjoyment, is also a strong predictor of PA participation, any intervention program should be designed to optimize their enjoyment of PA and thus enhance the likelihood of long-term adherence. When compared to structured exercises such as running or cycling, games-based PA arguably provides a more attractive, acceptable, sustainable, and enjoyable exercise model for young children. To date, only a few studies have examined the effect of an acute bout of team game-based activity on cognitive function in healthy children and adolescents. Research has found that different aspects of cognitive function, such as free recall memory, attention, executive function, and working memory are improved following an acute bout of game-based team exercise (e.g., basketball, tennis). For children with ADHD, mixed exercise protocols have generally been used in intervention programs, and only a few studies have used team sport-based games as part of their exercise intervention. However, given the design of these studies, it is not possible to distinguish the sole effect of game-based PA from those of the mixed exercise protocols in these studies. A recent study has reported that a 12-week table tennis exercise has positive effects on the gross motor skills and some of the executive function performances (mainly inhibition) in the ADHD training group, compared with the ADHD non-training group and a control group. It should be noted that the game-based PA in these aforementioned studies was generally 'aerobic' in nature and completed at low- to moderate intensities.

Recently high-intensity interval training (HIIT) has emerged as a feasible and efficacious strategy for improving the physical health of young people. The HIIT can be completed in a short period of time while resulting in equivalent physiological adaptations to longer sessions of traditional aerobic training. Recent research has suggested that traditional HIIT intervention programs, including running and cycling, may improve executive function in healthy children and adolescents. It has been suggested that a very brief HIIT intervention over two weeks reduced off-task behavior and enhanced selective attention in primary school children. For children with ADHD, to the best of our knowledge, only one recent study was conducted to investigate the effect of a traditional HIIT program on physical fitness, motor skills, social behavior, and quality of life. In this randomized controlled trial, 28 boys with ADHD were assigned to either a traditional HIIT group or a standard multimodal therapy (TRAD) group. After the three-week intervention, the authors reported that HIIT was more effective in improving motor skills, self-esteem, relations with friends, competence, and subjective ratings of attention, compared with TRAD. However, despite this encouraging preliminary evidence, it remains unclear whether HIIT can be adapted to treat children with ADHD to improve their executive function, a key aspect in many facets of life.

While the limited findings regarding the effects of HIIT on executive function are encouraging, and HIIT has emerged as an enjoyable and effective exercise for children, previous studies have tended to prescribe HIIT interventions with a focus on running and jumping. The effect of game-based HIIT interventions on the executive function of children has yet to be investigated. Research of this nature is needed, particularly to determine whether game-based HIIT can improve outcomes (e.g., executive function, social behavior, sports skills, etc.) for children with ADHD. Therefore, the aim of the proposed study is to investigate the effect of two different kinds of exercise programs, i.e., an 8-week game-based HIIT (GameHIIT) program and an 8-week game-based structured aerobic exercise (GameSAE) program, on the executive function of children with ADHD. The hypothesis of the proposed study is that both GameHIIT and GameSAE programs will significantly improve the executive function of children with ADHD, compared with those in the control group. A secondary hypothesis is that the GameHIIT group may confer additional benefits when compared with the GameSAE group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ADHD
* Must be able to participate in physical activity

Exclusion Criteria:

* Neurodevelopmental or psychiatric disorder (e.g., autism spectrum disorder, intellectual disability.
* Acute/chronic diseases that may affect engagement in physical activity
* A tendency to experience convulsions

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Colour-Word Stroop Test (CWST) | The measurements are assessed at baseline (T0).
  The executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Corsi Block Tapping Test (CBTT) | The measurements are assessed at baseline (T0).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Wisconsin Card Sorting Test (WCST) | The measurements are assessed at baseline (T0).
  The executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of the important components of executive function.
Tower of London Test (TLT) | The measurements are assessed at baseline (T0).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Colour-Word Stroop Test (CWST) | The measurements are assessed after the 8-week intervention period (T1).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Corsi Block Tapping Test (CBTT) | The measurements are assessed after the 8-week intervention period (T1).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Wisconsin Card Sorting Test (WCST) | The measurements are assessed after the 8-week intervention period (T1).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Tower of London Test (TLT) | The measurements are assessed after the 8-week intervention period (T1).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Colour-Word Stroop Test (CWST) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Corsi Block Tapping Test (CBTT) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Wisconsin Card Sorting Test (WCST) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Tower of London Test (TLT) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Executive function will be assessed using a battery of tests on a laptop computer that will take approximately five minutes to complete. The battery of tests include the Colour-Word Stroop Test (CWST), Corsi Block Tapping Test (CBTT), Wisconsin Card Sorting Test (WCST), and Tower of London Test (TLT) which are classic tasks that measure inhibition response, one of important components of executive function.
Cerebral Hemodynamic Response | The measurements are assessed at baseline (T0).
  Accompanied by the executive function test, the cortical hemodynamic response in the prefrontal cortex will also be recorded using a multi-channel fNIRS (Octamon fNIRS system, Artinis, Netherland) applying two wavelengths of near-infrared light (785 and 830 nm). The device consists of eight light sources and two detectors secured onto a head cap. The device will be placed over the left and right prefrontal cortex according to the guidelines in the handbook provided by the manufacturer.
Cerebral Hemodynamic Response | The measurements are assessed after the 8-week intervention period (T1).
  Accompanied by the executive function test, the cortical hemodynamic response in the prefrontal cortex will also be recorded using a multi-channel fNIRS (Octamon fNIRS system, Artinis, Netherland) applying two wavelengths of near-infrared light (785 and 830 nm). The device consists of eight light sources and two detectors secured onto a head cap. The device will be placed over the left and right prefrontal cortex according to the guidelines in the handbook provided by the manufacturer.
Cerebral Hemodynamic Response | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Accompanied by the executive function test, the cortical hemodynamic response in the prefrontal cortex will also be recorded using a multi-channel fNIRS (Octamon fNIRS system, Artinis, Netherland) applying two wavelengths of near-infrared light (785 and 830 nm). The device consists of eight light sources and two detectors secured onto a head cap. The device will be placed over the left and right prefrontal cortex according to the guidelines in the handbook provided by the manufacturer.

SECONDARY OUTCOMES:
Body height | The measurements are assessed at baseline (T0).
  Body height will be measured in meters. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Body height | The measurements are assessed after the 8-week intervention period (T1).
  Body height will be measured in meters. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Body height | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Body height will be measured in meters. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Body weight | The measurements are assessed at baseline (T0).
  Bodyweight will be measured in kilograms. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Body weight | The measurements are assessed after the 8-week intervention period (T1).
  Bodyweight will be measured in kilograms. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Body weight | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Bodyweight will be measured in kilograms. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES). Weight and height will be combined to report BMI in kg/m^2.
Waist circumference | The measurements are assessed at baseline (T0).
  Waist circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Waist circumference | The measurements are assessed after the 8-week intervention period (T1).
  Waist circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Waist circumference | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Waist circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Hip circumference | The measurements are assessed at baseline (T0).
  Hip circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Hip circumference | The measurements are assessed after the 8-week intervention period (T1).
  Hip circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Hip circumference | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Hip circumference will be measured and presented in centimetres. The measurement will follow the Anthropometry Procedures Manual of the National Health and Nutrition Examination Survey (NHANES).
Body mass index (BMI) | The measurements are assessed at baseline (T0).
  Weight and height will be combined to report BMI in kg/m^2.
Body mass index (BMI) | The measurements are assessed after the 8-week intervention period (T1).
  Weight and height will be combined to report BMI in kg/m^2.
Body mass index (BMI) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Weight and height will be combined to report BMI in kg/m^2.
Social Behavior | The measurements are assessed at baseline (T0).
  Conners' Teacher Rating Scale 15-Item (CTRS-15) will be used to measure the social behaviours of participants. It has been widely used to assess problematic behaviours in children with ADHD.
Social Behavior | The measurements are assessed after the 8-week intervention period (T1).
  Conners' Teacher Rating Scale 15-Item (CTRS-15) will be used to measure the social behaviours of participants. It has been widely used to assess problematic behaviours in children with ADHD.
Social Behavior | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Conners' Teacher Rating Scale 15-Item (CTRS-15) will be used to measure the social behaviours of participants. It has been widely used to assess problematic behaviours in children with ADHD.
Overall ADHD Symptoms | The measurements are assessed at baseline (T0).
  The Overall ADHD symptoms will be assessed by the Attention-Deficit/Hyperactivity-symptoms and Normal-behaviors (SWAN) rating scale (0-3), the scale scores in '0' means 'Not true' and '3' in 'Very much true'.
Overall ADHD Symptoms | The measurements are assessed after the 8-week intervention period (T1).
  The Overall ADHD symptoms will be assessed by the Attention-Deficit/Hyperactivity-symptoms and Normal-behaviors (SWAN) rating scale (0-3), the scale scores in '0' means 'Not true' and '3' in 'Very much true'.
Overall ADHD Symptoms | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  The Overall ADHD symptoms will be assessed by the Attention-Deficit/Hyperactivity-symptoms and Normal-behaviors (SWAN) rating scale (0-3), the scale scores in '0' means 'Not true' and '3' in 'Very much true'.
Moderate-to-Vigorous Physical Activity (MVPA) | The measurements are assessed at baseline (T0).
  Children's leisure-time MVPA will be determined using an accelerometer (ActiGraph, Shalimar, USA).Participants will be required to wear an accelerometer on their right hip for seven days to collect objective data of PA levels. The time on and time off of wearing the accelerometer each day will be recorded, and the data will be used to estimate the time spent in moderate-to-vigorous PA (MVPA).
Moderate-to-Vigorous Physical Activity (MVPA) | The measurements are assessed after the 8-week intervention period (T1).
  Children's leisure-time MVPA will be determined using an accelerometer (ActiGraph, Shalimar, USA).Participants will be required to wear an accelerometer on their right hip for seven days to collect objective data of PA levels. The time on and time off of wearing the accelerometer each day will be recorded, and the data will be used to estimate the time spent in moderate-to-vigorous PA (MVPA).
Moderate-to-Vigorous Physical Activity (MVPA) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Children's leisure-time MVPA will be determined using an accelerometer (ActiGraph, Shalimar, USA).Participants will be required to wear an accelerometer on their right hip for seven days to collect objective data of PA levels. The time on and time off of wearing the accelerometer each day will be recorded, and the data will be used to estimate the time spent in moderate-to-vigorous PA (MVPA).
Self-reported Physical Activity | The measurements are assessed at baseline (T0).
  The modified version of the Physical Activity Questionnaire for Children (PAQ-C) is a 7-day self-report questionnaire designed to assess daily activities from moderate to the vigorous range, and the score is in a continuous range from 1 (low active) to 5 (high active).
Self-reported Physical Activity | The measurements are assessed after the 8-week intervention period (T1).
  The modified version of the Physical Activity Questionnaire for Children (PAQ-C) is a 7-day self-report questionnaire designed to assess daily activities from moderate to the vigorous range, and the score is in a continuous range from 1 (low active) to 5 (high active).
Self-reported Physical Activity | The measurements are assessed after the 8-week intervention period and another 8-week follow up (T2).
  The modified version of the Physical Activity Questionnaire for Children (PAQ-C) is a 7-day self-report questionnaire designed to assess daily activities from moderate to the vigorous range, and the score is in a continuous range from 1 (low active) to 5 (high active).
Enjoyment | The measurements are assessed at baseline (T0).
  Enjoyment will be assessed by the Physical Activity Enjoyment Scale, which is a valid and reliable tool for evaluating perceived enjoyment. The PACES consisted of 18 bipolar statements on a 7-point continuum (I enjoy it-I hate it) which are summed to produce a total enjoyment score.
Enjoyment | The measurements are assessed after the 8-week intervention period (T1).
  Enjoyment will be assessed by the Physical Activity Enjoyment Scale, which is a valid and reliable tool for evaluating perceived enjoyment. The PACES consisted of 18 bipolar statements on a 7-point continuum (I enjoy it-I hate it) which are summed to produce a total enjoyment score.
Enjoyment | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Enjoyment will be assessed by the Physical Activity Enjoyment Scale, which is a valid and reliable tool for evaluating perceived enjoyment. The PACES consisted of 18 bipolar statements on a 7-point continuum (I enjoy it-I hate it) which are summed to produce a total enjoyment score.
Adherence | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  Adherence to the intervention program will be evaluated by attendance frequency and dropout rate.
Physical Fitness (cardiovascular fitness) | The measurements are assessed at baseline (T0).
  The cardiovascular fitness will be assessed by the 20 m shuttle run test using the ALPHA fitness test battery.
Physical Fitness (cardiovascular fitness) | The measurements are assessed after the 8-week intervention period (T1).
  The cardiovascular fitness will be assessed by the 20 m shuttle run test using the ALPHA fitness test battery.
Physical Fitness (cardiovascular fitness) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  The cardiovascular fitness will be assessed by the 20 m shuttle run test using the ALPHA fitness test battery.
Physical Fitness (muscular strength) | The measurements are assessed at baseline (T0).
  The muscular strength will be assessed by the handgrip strength test and standing long jump test using the ALPHA fitness test battery.
Physical Fitness (muscular strength) | The measurements are assessed after the 8-week intervention period (T1).
  The muscular strength will be assessed by the handgrip strength test and standing long jump test using the ALPHA fitness test battery.
Physical Fitness (muscular strength) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  The muscular strength will be assessed by the handgrip strength test and standing long jump test using the ALPHA fitness test battery.
Physical Fitness (speed-agility) | The measurements are assessed at baseline (T0).
  The speed-agility will be assessed by the 4 × 10 m shuttle run test using the ALPHA fitness test battery.
Physical Fitness (speed-agility) | The measurements are assessed after the 8-week intervention period (T1).
  The speed-agility will be assessed by the 4 × 10 m shuttle run test using the ALPHA fitness test battery.
Physical Fitness (speed-agility) | The measurements are assessed after the 8-week intervention period, as well as another 8-week follow up (T2).
  The speed-agility will be assessed by the 4 × 10 m shuttle run test using the ALPHA fitness test battery.

CONTACTS AND LOCATIONS:
Overall Officials: Fenghua Sun, Dotcor, Study Director — The Education University of Hong Kong
Locations (1):
- The Education University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janssen I, Leblanc AG. Systematic review of the health benefits of physical activity and fitness in school-aged children and youth. Int J Behav Nutr Phys Act. 2010 May 11;7:40. doi: 10.1186/1479-5868-7-40. PMID 20459784
- [Background] Parfitt G, Eston RG. The relationship between children's habitual activity level and psychological well-being. Acta Paediatr. 2005 Dec;94(12):1791-7. doi: 10.1111/j.1651-2227.2005.tb01855.x. PMID 16421041
- [Background] Hillman CH, Erickson KI, Kramer AF. Be smart, exercise your heart: exercise effects on brain and cognition. Nat Rev Neurosci. 2008 Jan;9(1):58-65. doi: 10.1038/nrn2298. PMID 18094706
- [Background] Alvarez JA, Emory E. Executive function and the frontal lobes: a meta-analytic review. Neuropsychol Rev. 2006 Mar;16(1):17-42. doi: 10.1007/s11065-006-9002-x. PMID 16794878
- [Background] Kramer AF, Humphrey DG, Larish JF, Logan GD, Strayer DL. Aging and inhibition: beyond a unitary view of inhibitory processing in attention. Psychol Aging. 1994 Dec;9(4):491-512. PMID 7893421
- [Background] Pennington BF, Ozonoff S. Executive functions and developmental psychopathology. J Child Psychol Psychiatry. 1996 Jan;37(1):51-87. doi: 10.1111/j.1469-7610.1996.tb01380.x. PMID 8655658
- [Background] Diamond A. Executive functions. Annu Rev Psychol. 2013;64:135-68. doi: 10.1146/annurev-psych-113011-143750. Epub 2012 Sep 27. PMID 23020641
- [Background] Moffitt TE, Arseneault L, Belsky D, Dickson N, Hancox RJ, Harrington H, Houts R, Poulton R, Roberts BW, Ross S, Sears MR, Thomson WM, Caspi A. A gradient of childhood self-control predicts health, wealth, and public safety. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):2693-8. doi: 10.1073/pnas.1010076108. Epub 2011 Jan 24. PMID 21262822
- [Background] Verburgh L, Konigs M, Scherder EJ, Oosterlaan J. Physical exercise and executive functions in preadolescent children, adolescents and young adults: a meta-analysis. Br J Sports Med. 2014 Jun;48(12):973-9. doi: 10.1136/bjsports-2012-091441. Epub 2013 Mar 6. PMID 23467962
- [Background] Alvarez-Bueno C, Pesce C, Cavero-Redondo I, Sanchez-Lopez M, Martinez-Hortelano JA, Martinez-Vizcaino V. The Effect of Physical Activity Interventions on Children's Cognition and Metacognition: A Systematic Review and Meta-Analysis. J Am Acad Child Adolesc Psychiatry. 2017 Sep;56(9):729-738. doi: 10.1016/j.jaac.2017.06.012. Epub 2017 Jul 6. PMID 28838577
- [Background] Huang WY, Wong SHS, Sit CHP, Wong MCS, Sum RKW, Wong SWS, Yu JJ. Results from the Hong Kong's 2018 report card on physical activity for children and youth. J Exerc Sci Fit. 2019 Jan;17(1):14-19. doi: 10.1016/j.jesf.2018.10.003. Epub 2018 Oct 8. PMID 30662509
- [Background] Mak KK, Day JR. Secular trends of sports participation, sedentary activity and physical self-perceptions in Hong Kong adolescents, 1995-2000. Acta Paediatr. 2010 Nov;99(11):1731-4. doi: 10.1111/j.1651-2227.2010.01928.x. Epub 2010 Jul 13. PMID 20586996
- [Background] Blakemore SJ, Choudhury S. Development of the adolescent brain: implications for executive function and social cognition. J Child Psychol Psychiatry. 2006 Mar-Apr;47(3-4):296-312. doi: 10.1111/j.1469-7610.2006.01611.x. PMID 16492261
- [Background] Zelazo PD, Craik FI, Booth L. Executive function across the life span. Acta Psychol (Amst). 2004 Feb-Mar;115(2-3):167-83. doi: 10.1016/j.actpsy.2003.12.005. PMID 14962399
- [Background] Best JR, Miller PH, Jones LL. Executive Functions after Age 5: Changes and Correlates. Dev Rev. 2009 Sep 1;29(3):180-200. doi: 10.1016/j.dr.2009.05.002. PMID 20161467
- [Background] Cotman CW, Berchtold NC. Exercise: a behavioral intervention to enhance brain health and plasticity. Trends Neurosci. 2002 Jun;25(6):295-301. doi: 10.1016/s0166-2236(02)02143-4. PMID 12086747
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Barkley RA. Adolescents with attention-deficit/hyperactivity disorder: an overview of empirically based treatments. J Psychiatr Pract. 2004 Jan;10(1):39-56. doi: 10.1097/00131746-200401000-00005. PMID 15334986
- [Background] Ng QX, Ho CYX, Chan HW, Yong BZJ, Yeo WS. Managing childhood and adolescent attention-deficit/hyperactivity disorder (ADHD) with exercise: A systematic review. Complement Ther Med. 2017 Oct;34:123-128. doi: 10.1016/j.ctim.2017.08.018. Epub 2017 Aug 31. PMID 28917364
- [Background] Neudecker C, Mewes N, Reimers AK, Woll A. Exercise Interventions in Children and Adolescents With ADHD: A Systematic Review. J Atten Disord. 2019 Feb;23(4):307-324. doi: 10.1177/1087054715584053. Epub 2015 May 11. PMID 25964449
- [Background] Den Heijer AE, Groen Y, Tucha L, Fuermaier AB, Koerts J, Lange KW, Thome J, Tucha O. Sweat it out? The effects of physical exercise on cognition and behavior in children and adults with ADHD: a systematic literature review. J Neural Transm (Vienna). 2017 Feb;124(Suppl 1):3-26. doi: 10.1007/s00702-016-1593-7. Epub 2016 Jul 11. PMID 27400928
- [Background] Chang YK, Liu S, Yu HH, Lee YH. Effect of acute exercise on executive function in children with attention deficit hyperactivity disorder. Arch Clin Neuropsychol. 2012 Mar;27(2):225-37. doi: 10.1093/arclin/acr094. Epub 2012 Feb 3. PMID 22306962
- [Background] Pontifex MB, Saliba BJ, Raine LB, Picchietti DL, Hillman CH. Exercise improves behavioral, neurocognitive, and scholastic performance in children with attention-deficit/hyperactivity disorder. J Pediatr. 2013 Mar;162(3):543-51. doi: 10.1016/j.jpeds.2012.08.036. Epub 2012 Oct 17. PMID 23084704
- [Background] Chang YK, Hung CL, Huang CJ, Hatfield BD, Hung TM. Effects of an aquatic exercise program on inhibitory control in children with ADHD: a preliminary study. Arch Clin Neuropsychol. 2014 May;29(3):217-23. doi: 10.1093/arclin/acu003. Epub 2014 Apr 2. PMID 24695590
- [Background] Choi JW, Han DH, Kang KD, Jung HY, Renshaw PF. Aerobic exercise and attention deficit hyperactivity disorder: brain research. Med Sci Sports Exerc. 2015 Jan;47(1):33-9. doi: 10.1249/MSS.0000000000000373. PMID 24824770
- [Background] Verret C, Guay MC, Berthiaume C, Gardiner P, Beliveau L. A physical activity program improves behavior and cognitive functions in children with ADHD: an exploratory study. J Atten Disord. 2012 Jan;16(1):71-80. doi: 10.1177/1087054710379735. Epub 2010 Sep 13. PMID 20837978
- [Background] Banaschewski T, Besmens F, Zieger H, Rothenberger A. Evaluation of sensorimotor training in children with ADHD. Percept Mot Skills. 2001 Feb;92(1):137-49. doi: 10.2466/pms.2001.92.1.137. PMID 11322578
- [Background] Biddle SJ, Gorely T, Stensel DJ. Health-enhancing physical activity and sedentary behaviour in children and adolescents. J Sports Sci. 2004 Aug;22(8):679-701. doi: 10.1080/02640410410001712412. PMID 15370482
- [Background] Nassis GP, Papantakou K, Skenderi K, Triandafillopoulou M, Kavouras SA, Yannakoulia M, Chrousos GP, Sidossis LS. Aerobic exercise training improves insulin sensitivity without changes in body weight, body fat, adiponectin, and inflammatory markers in overweight and obese girls. Metabolism. 2005 Nov;54(11):1472-9. doi: 10.1016/j.metabol.2005.05.013. PMID 16253636
- [Background] Sebire SJ, Jago R, Fox KR, Edwards MJ, Thompson JL. Testing a self-determination theory model of children's physical activity motivation: a cross-sectional study. Int J Behav Nutr Phys Act. 2013 Sep 26;10:111. doi: 10.1186/1479-5868-10-111. PMID 24067078
- [Background] Cooper SB, Dring KJ, Nevill ME. High-Intensity Intermittent Exercise: Effect on Young People's Cardiometabolic Health and Cognition. Curr Sports Med Rep. 2016 Jul-Aug;15(4):245-51. doi: 10.1249/JSR.0000000000000273. PMID 27399821
- [Background] Cooper SB, Dring KJ, Morris JG, Sunderland C, Bandelow S, Nevill ME. High intensity intermittent games-based activity and adolescents' cognition: moderating effect of physical fitness. BMC Public Health. 2018 May 8;18(1):603. doi: 10.1186/s12889-018-5514-6. PMID 29739386
- [Background] Ishihara T, Sugasawa S, Matsuda Y, Mizuno M. The beneficial effects of game-based exercise using age-appropriate tennis lessons on the executive functions of 6-12-year-old children. Neurosci Lett. 2017 Mar 6;642:97-101. doi: 10.1016/j.neulet.2017.01.057. Epub 2017 Jan 31. PMID 28159634
- [Background] Gallotta MC, Guidetti L, Franciosi E, Emerenziani GP, Bonavolonta V, Baldari C. Effects of varying type of exertion on children's attention capacity. Med Sci Sports Exerc. 2012 Mar;44(3):550-5. doi: 10.1249/MSS.0b013e3182305552. PMID 21814148
- [Background] Pan CY, Tsai CL, Chu CH, Sung MC, Huang CY, Ma WY. Effects of Physical Exercise Intervention on Motor Skills and Executive Functions in Children With ADHD: A Pilot Study. J Atten Disord. 2019 Feb;23(4):384-397. doi: 10.1177/1087054715569282. Epub 2015 Feb 2. PMID 25646023
- [Background] Costigan SA, Eather N, Plotnikoff RC, Taaffe DR, Lubans DR. High-intensity interval training for improving health-related fitness in adolescents: a systematic review and meta-analysis. Br J Sports Med. 2015 Oct;49(19):1253-61. doi: 10.1136/bjsports-2014-094490. Epub 2015 Jun 18. PMID 26089322
- [Background] Logan GR, Harris N, Duncan S, Schofield G. A review of adolescent high-intensity interval training. Sports Med. 2014 Aug;44(8):1071-85. doi: 10.1007/s40279-014-0187-5. PMID 24743929
- [Background] Buchheit M, Laursen PB. High-intensity interval training, solutions to the programming puzzle: Part I: cardiopulmonary emphasis. Sports Med. 2013 May;43(5):313-38. doi: 10.1007/s40279-013-0029-x. PMID 23539308
- [Background] Ma JK, Le Mare L, Gurd BJ. Four minutes of in-class high-intensity interval activity improves selective attention in 9- to 11-year olds. Appl Physiol Nutr Metab. 2015 Mar;40(3):238-44. doi: 10.1139/apnm-2014-0309. Epub 2014 Nov 10. PMID 25675352
- [Background] Ma JK, Le Mare L, Gurd BJ. Classroom-based high-intensity interval activity improves off-task behaviour in primary school students. Appl Physiol Nutr Metab. 2014 Dec;39(12):1332-7. doi: 10.1139/apnm-2014-0125. Epub 2014 Jul 28. PMID 25263695
- [Background] Costigan SA, Eather N, Plotnikoff RC, Hillman CH, Lubans DR. High-Intensity Interval Training for Cognitive and Mental Health in Adolescents. Med Sci Sports Exerc. 2016 Oct;48(10):1985-93. doi: 10.1249/MSS.0000000000000993. PMID 27187097
- [Background] Messler CF, Holmberg HC, Sperlich B. Multimodal Therapy Involving High-Intensity Interval Training Improves the Physical Fitness, Motor Skills, Social Behavior, and Quality of Life of Boys With ADHD: A Randomized Controlled Study. J Atten Disord. 2018 Jun;22(8):806-812. doi: 10.1177/1087054716636936. Epub 2016 Mar 24. PMID 27013028
- [Background] Wigal SB, Emmerson N, Gehricke JG, Galassetti P. Exercise: applications to childhood ADHD. J Atten Disord. 2013 May;17(4):279-90. doi: 10.1177/1087054712454192. Epub 2012 Aug 3. PMID 22863768
- [Background] Anderson P. Assessment and development of executive function (EF) during childhood. Child Neuropsychol. 2002 Jun;8(2):71-82. doi: 10.1076/chin.8.2.71.8724. PMID 12638061
- [Background] Gary RA, Brunn K. Aerobic exercise as an adjunct therapy for improving cognitive function in heart failure. Cardiol Res Pract. 2014;2014:157508. doi: 10.1155/2014/157508. Epub 2014 Jul 3. PMID 25105053